CLINICAL TRIAL: NCT06378684
Title: A Randomized, Open-label, Multiple-dose, 6×3 Crossover Clinical Trial to Investigate the Pharmacokinetic Drug Interaction and Safety of JW0104 and C2207 in Healthy Adults
Brief Title: To Evaluate the Safety and Pharmacokinetic Interactions in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: JW22105
Record Dates: First submitted 2024-03-29; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 (Other): Treatment A: administration of 1 tablet of JW0104 Treatment B: administration of 1 tablet of C2207 Treatment A+B: Co-administration of 2 tablets of JW0104 and C2207
  Tablet, Oral, QD for 10 Days, Washout period is more than 14 days after administration
  Interventions: Drug: Group 1: JW0104(Period 1), C2207(Period 2), JW0104 + C2207(Period 3)
- Group 2 (Other): Treatment A: administration of 1 tablet of JW0104 Treatment B: administration of 1 tablet of C2207 Treatment A+B: Co-administration of 2 tablets of JW0104 and C2207
  Tablet, Oral, QD for 10 Days, Washout period is more than 14 days after administration
  Interventions: Drug: Group 2: JW0104 + C2207(Period 1), JW0104(Period 2), C2207(Period 3)
- Group 3 (Other): Treatment A: administration of 1 tablet of JW0104 Treatment B: administration of 1 tablet of C2207 Treatment A+B: Co-administration of 2 tablets of JW0104 and C2207
  Tablet, Oral, QD for 10 Days, Washout period is more than 14 days after administration
  Interventions: Drug: Group 3: C2207(Period 1), JW0104 + C2207(Period 2), JW0104(Period 3)
- Group 4 (Other): Treatment A: administration of 1 tablet of JW0104 Treatment B: administration of 1 tablet of C2207 Treatment A+B: Co-administration of 2 tablets of JW0104 and C2207
  Tablet, Oral, QD for 10 Days, Washout period is more than 14 days after administration
  Interventions: Drug: Group 4: JW0104(Period 1), JW0104 + C2207(Period 2), C2207(Period 3)
- Group 5 (Other): Treatment A: administration of 1 tablet of JW0104 Treatment B: administration of 1 tablet of C2207 Treatment A+B: Co-administration of 2 tablets of JW0104 and C2207
  Tablet, Oral, QD for 10 Days, Washout period is more than 14 days after administration
  Interventions: Drug: Group 5: JW0104 + C2207(Period 1), C2207(Period 2), JW0104(Period 3)
- Group 6 (Other): Treatment A: administration of 1 tablet of JW0104 Treatment B: administration of 1 tablet of C2207 Treatment A+B: Co-administration of 2 tablets of JW0104 and C2207
  Tablet, Oral, QD for 10 Days, Washout period is more than 14 days after administration
  Interventions: Drug: Group 6: C2207(Period 1), JW0104(Period 2), JW0104 + C2207(Period 3)

INTERVENTIONS:
Drug: Group 1: JW0104(Period 1), C2207(Period 2), JW0104 + C2207(Period 3) — Tablet, Oral, QD for 10 Days, Washout period is more than 14 days after administration
  Arms: Group 1
Drug: Group 2: JW0104 + C2207(Period 1), JW0104(Period 2), C2207(Period 3) — Tablet, Oral, QD for 10 Days, Washout period is more than 14 days after administration
  Arms: Group 2
Drug: Group 3: C2207(Period 1), JW0104 + C2207(Period 2), JW0104(Period 3) — Tablet, Oral, QD for 10 Days, Washout period is more than 14 days after administration
  Arms: Group 3
Drug: Group 4: JW0104(Period 1), JW0104 + C2207(Period 2), C2207(Period 3) — Tablet, Oral, QD for 10 Days, Washout period is more than 14 days after administration
  Arms: Group 4
Drug: Group 5: JW0104 + C2207(Period 1), C2207(Period 2), JW0104(Period 3) — Tablet, Oral, QD for 10 Days, Washout period is more than 14 days after administration
  Arms: Group 5
Drug: Group 6: C2207(Period 1), JW0104(Period 2), JW0104 + C2207(Period 3) — Tablet, Oral, QD for 10 Days, Washout period is more than 14 days after administration
  Arms: Group 6

SUMMARY:
The objective is to evaluate the safety and Pharmacokinetic Interactions after adminitration drug(Treatment A or B or A+B) in Healthy Volunteers

DETAILED DESCRIPTION:
Pharmacokinetic Interactions: Describes the blood concentration statistically by pharmacokinetic blood collection time and treatment group.

Safety: All adverse events are summarized in terms of the number of subjects, expression rate, and number of expressions of adverse reactions by treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Subjects does not meet the Inclusion Criteria

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-09-10 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2024-01-13 (Actual)

PRIMARY OUTCOMES:
Cmax,ss | Day 1(0 hour), Day 8(0 hour), Day 9(0 hour), Day 10(0 hour) ~ Day 13(72 hours)
  Describes the blood concentration statistically by pharmacokinetic blood collection time and treatment group.
AUCτ,ss | Day 1(0 hour), Day 8(0 hour), Day 9(0 hour), Day 10(0 hour) ~ Day 13(72 hours)
  Describes the blood concentration statistically by pharmacokinetic blood collection time and treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: MinSoo Kim, Principal Investigator — Severance Hospital
Locations (1):
- Clinical Trial Center, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No